CLINICAL TRIAL: NCT02553837
Title: Study to Evaluate the Immunogenicity and Safety of Hantavax in Healthy Adult
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GC3101B_P3
Record Dates: First submitted 2015-09-13; First posted 2015-09-18 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment only (Experimental): Drug: Hantavax injectionSchedule: The basic vaccination(0, 1, 2months) and The boost vaccination(13months)
  Interventions: Biological: Hantavax injection

INTERVENTIONS:
Biological: Hantavax injection — A single 0.5mL dose intramuscular or subcutaneous injection

SUMMARY:
This study was aimed to evaluate the Immunogenicity and Safety response by vaccinating Hantavax in Healthy Adult.

DETAILED DESCRIPTION:
This clinical trial was designed as a multicenter, non-comparative, open-label clinical trial. This trial was conducted, written informed consent form by voluntary agreement, the subjects who have not had the hantavax vaccination history at the time of screening. Investigator product was administrated 0, 1, 2, 13 months.

For antibody test, Sampling was conducted pre-dose(T0), 28 days after the 2nd vaccination(before the 3rd vaccination, T1), 28 days after the 3rd vaccination(T2) and 11 months after the 3rd vaccination(before booster vaccination, T3), 28 days after the booster vaccination(T4), 2 months after the booster vaccination(T5) and 4 months after the booster vaccination(T6). Also, after the completion of booster vaccination for antibody retention duration observed for subjects with antibody to conduct a five-year follow-up survey was conducted, and the antibody test every year. In conclusion, sampling was conducted 12 months(T7), 24 months(T8), 36months(T9), 48 months(T10), 60 months(T11) after the booster vaccination.

However, follow-up survey was terminated when the antibody titer was determined as a negative by neutralizing antibody test and fluorescent antibody technique.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ≥ 19years old.
* Subjects who have not the hantavax vaccination history at the time of screening.

Exclusion Criteria:

* Subject who did not passed by 2 weeks after recovering the acute disease.
* immunologic dysfunction subjects.
* Subjects previously treated with anti-coagulant therapy or hemophiliac patients.
* Subjects with severe chronic diseases.
* Subjects who had an acute before vaccinating IP.
* Subjects who had received another vaccination during the 28 days before vaccinating IP or who were scheduled for another vaccination during the study.
* Subjects who were receiving immunosuppressant or immune modifying drug
* Subjects who had been administered immunoglobulins or blood-derived products 3 months before vaccinating IP or who were scheduled for the administration during the study.
* Subjects of childbearing potential at the time of screening and were scheduled to pregnancy for the study. A female subject who was pregnant or who was breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 317 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-08 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
The Antibody Seroconversion rates by neutralizing antibody test at 28 days after the 3rd vaccination(2month) | 3 months

SECONDARY OUTCOMES:
The Antibody Seroconversion Rates by fluorescent antibody test at 28 days after the 3rd vaccination(2month) | 3 months
The Antibody Seroconversion Rates by neutralizing antibody test and fluorescent antibody test at 28 days after the 2nd vaccination(1month) | 2 months
The Antibody Seroconversion Rates by neutralizing antibody test and fluorescent antibody test at 28 days after the 4th vaccination(13month) | 14 months
The Antibody Seroconversion Rates by neutralizing antibody test and fluorescent antibody test at 2 , 4, 12, 24, 36, 48, 60months after the 4th vaccination(13month) | 15, 17, 25, 37, 49, 61, 73months
Geometric Mean Titer(GMT) at 28 days after the 2nd vaccination(1month) | 2 months
Geometric Mean Titer(GMT) at 28 days after the 3rd vaccination(2month) | 3 months
Geometric Mean Titer(GMT) at 28 days after the 4th vaccination(13month) | 14 months
Geometric Mean Titer(GMT) at 2, 4, 12, 24, 36, 48, 60 after the 4th vaccination(13month) | 15, 17, 25, 37, 49, 61, 73months
The Antibodies retention duration per the neutralizing antibody test | 5 years
The Antibodies retention duration per the fluorescent antibody test | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo Kim, MD, Principal Investigator — Korea University Guro Hospital

REFERENCES:
- [Derived] Song JY, Jeong HW, Yun JW, Lee J, Woo HJ, Bae JY, Park MS, Choi WS, Park DW, Noh JY, Cheong HJ, Kim WJ. Immunogenicity and safety of a modified three-dose priming and booster schedule for the Hantaan virus vaccine (Hantavax): A multi-center phase III clinical trial in healthy adults. Vaccine. 2020 Nov 25;38(50):8016-8023. doi: 10.1016/j.vaccine.2020.10.035. Epub 2020 Oct 31. PMID 33131933